CLINICAL TRIAL: NCT00927875
Title: A Phase 1b Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-833923 (XL139) in Combination With Carboplatin and Etoposide Followed by BMS-833923 Alone in Subjects With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of BMS-833923 With Carboplatin and Etoposide Followed by BMS-833923 Alone in Subjects With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA194-005; 2010-018745-56 (EudraCT Number)
Record Dates: First submitted 2009-06-09; First posted 2009-06-25 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — BMS-833923; Carboplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental)
  Interventions: Drug: BMS-833923; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: BMS-833923 — Capsule, Oral, starting dose 30 mg, once daily, continuous
Drug: Carboplatin — Vial, Intravenous (IV), dose to yield 5 mg/mL - min, once every 21 days, 1 day per cycle up to 4 cycles
  Other Names: Paraplatin®
Drug: Etoposide — Vial, Intravenous (IV), 100 mg/m²/dose, days 1, 2, & 3 of each 21 day cycle, 3 days per cycle for up to 4 cycles
  Other Names: Etopophos®; Toposar®; VePesid®

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of BMS-833923 administered in combination with carboplatin and etoposide followed by BMS-833923 alone in subjects with extensive-stage Small Cell Lung Cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer, without prior chemotherapy treatment
* Men and Women at least 18 years old
* Eastern Cooperative Oncology Group (ECOG) status 0-2

Exclusion Criteria:

* Significant cardiovascular disease
* Prior treatment of small cell lung cancer is not permitted, except for palliative radiation to a limited field excluding the chest (e.g. for painful metastasis).
* Symptomatic brain metastases
* Women pregnant or breastfeeding
* Women of childbearing potential (WOCBP) unwilling/unable to use acceptable method to avoid pregnancy
* Uncontrolled medical disorder or active infection
* Concurrent therapy with any other investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Use NCI CTCAE to establish the MTD, DLT(s) and safety profile of BMS-833923 administered alone and in combination with carboplatin and etoposide | 28 days
  * NCI - National Cancer Institute
  * CTCAE - Common Terminology Criteria for Adverse Events
  * MTD - Maximum tolerated dose
  * DLT - Dose limiting toxicity

SECONDARY OUTCOMES:
Pharmacokinetic parameters of BMS-833923 alone and in combination with carboplatin and etoposide: Maximum observed plasma concentration (Cmax) | Day 1 and 15 of first three 21-day cycles
Pharmacokinetic parameters of BMS-833923 alone and in combination with carboplatin and etoposide: Time of maximum observed plasma concentration (Tmax) | Day 1 and 15 of first three 21-day cycles
Pharmacokinetic parameters of BMS-833923 alone and in combination with carboplatin and etoposide: Area under the concentration-time curve in one dosing interval AUC(TAU) | Day 1 and 15 of first three 21-day cycles
Tumor assessments by computed tomography (CT) [as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1] | Every 6 weeks until disease progression
Pharmacodynamic effect (change from baseline) of BMS-833923 on Hedgehog pathway activation as measured by Glioma-associated oncogene -1 (GLI-1) expression | At baseline and after 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Karmanos Cancer Institute, Detroit, Michigan, United States
- Local Institution, East Bentleigh, Victoria, Australia
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
- Local Institution, Villejuif, France
- Local Institution, Dublin, Dublin, Ireland

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx